CLINICAL TRIAL: NCT05652166
Title: What Information is Remembered by Parents Following the Ingestion of Foreign Body by Their Child?
Acronym: MICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP-MICE
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-11

CONDITIONS: Information Remembered by Parents Following the Ingestion of Foreign Body by Their Child
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: telephone interview — telephone call to parents to know the information given following the ingestion of foreign body by their child

SUMMARY:
Foreign body (FB) ingestion is a very common domestic accident in children. The prevention of the recurrence by securing child's environment is mandatory. The study will study whether the advices of follow-up at home and recurrence prophylaxis were given to parents after a foreign ingestion by their child.

DETAILED DESCRIPTION:
Foreign body ingestion (FB) is a very common domestic accident in children. When the FB is not dangerous or it is inaccessible after crossing the pylorus, the child should be monitored. In all cases, recurrence should be prevented by securing the environment of the swallowing child. The information on monitoring and securing the environment should be communicated during hospital care. This prospective study will analyze whether advices were correctly given to the families concerning the follow-up at home and the prophylaxis of FB ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Children under 18 years
* Foreign body ingestion

Exclusion Criteria:

* Refusal to participate in the study
* Non-French speaking parents

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children consulting at Robert Debre Hospital following the ingestion of foreign body
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Identify the instructions memorized by the parents after a visit to the hospital for a foreign body ingestion by their child. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme VIALA, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided